CLINICAL TRIAL: NCT05408533
Title: Silver-coated Catheter Versus Standard Catheter for UTI Prevention in a Short-term Transurethral Indwelling Catheter Population After Pelvic Reconstructive Surgery: A Randomized Controlled Trial
Brief Title: Silver-Coated vs Standard Catheter for UTI Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 22-004
Record Dates: First submitted 2022-04-29; First posted 2022-06-07 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: UTI
Keywords: Silver-coated catheter; UTI; Pelvic Reconstructive Surgery; Urogynecology

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Silver-Coated Catheter (Active Comparator)
  Interventions: Device: 2-Way Foley Urethral Urinary Catheter
- Standard Catheter (Placebo Comparator)
  Interventions: Device: 2-Way Foley Urethral Urinary Catheter

INTERVENTIONS:
Device: 2-Way Foley Urethral Urinary Catheter — Comparing two types of catheter (silver-coated silicone versus silicone) after Pelvic Reconstructive Surgery (PRS) to compare Urinary Tract Infection (UTI) rates

SUMMARY:
Primary Aim: To determine whether silver-coated transurethral catheter decreases the incidence of culture-confirmed urinary tract infection for women with catheter-managed urinary retention after pelvic reconstructive surgery

Secondary Aims:

To assess difference in bacterial uropathogens isolated in urine cultures Adverse symptoms possibly caused by silver-coated catheter

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo major or minor pelvic organ prolapse surgery of any compartment, or urinary incontinence surgery that are diagnosed with POUR via failed retrograde voiding trial and require an indwelling transurethral catheter upon hospital discharge. Sacral neuromodulation procedures and intradetrusor onabotulinumtoxinA (Botox) injections are excluded.

Exclusion Criteria:

* Unwilling or unable to participate in the study.
* Unwilling or unable to do a catheter self-removal at home.
* Inability to understand English.
* Pregnant women
* Patient personal history of urogenital anomaly, neurogenic bladder, use of chronic self-intermittent catheterization or suprapubic tubes, ureteral stents or other genitourinary indwelling devices, immunosuppressed state or chronic use of steroids.
* Currently (prior 3 months) undergoing medical management for recurrent UTI or interstitial cystitis
* Active urinary tract infection.
* Intraoperative bladder injury or cystotomy
* Physical or mental impairment that would affect the subject's ability to perceive urinary tract infection symptoms
* Reported allergy to silver metal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of UTIs requiring treatment | approximately 4 weeks
  Post-operative UTI rate

SECONDARY OUTCOMES:
Assess the types of bacterial uropathogens isolated from the urine cultures | approximately 4 weeks
Adverse symptoms possibly causes by silver-coated catheter | approximately 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Yeung, DO, Principal Investigator — TriHealth Inc.
Locations (2):
- United States (2):
  - Cincinnati Urogynecology Associates, Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lewis K, Crisp C, Ray M, Bonglack M, Carrel-Lammert M, Aldrich E, Pauls R, Hoehn J, Yeung J. Silver-Coated Foley Catheters to Reduce UTIs: A Randomized Clinical Trial. Urogynecology (Phila). 2025 Mar 1;31(3):276-284. doi: 10.1097/SPV.0000000000001634. Epub 2025 Jan 2. PMID 39744866